CLINICAL TRIAL: NCT00403845
Title: A Randomized, Double-blind, Placebo-controlled, 4-period 4-treatment Crossover, Multicenter, Dose-ranging Study to Assess the Efficacy and Safety of 3 Doses of Indacaterol (150, 300, and 600 µg) Delivered Via a Single Dose Dry Powder Inhaler in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Dose Ranging Study of Indacaterol in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B1202
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; QAB149; indacaterol; long acting β2-agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo-indacaterol 150μg-indacaterol 300μg-indacaterol 600μg (Experimental): In treatment period, 1 patients received 2 placebo capsules; in treatment period 2, patients received 1 indacaterol 150 μg capsule + 1 placebo capsule; in treatment period 3, patients received 1 indacaterol 300 μg capsule + 1 placebo capsule; and in treatment period 4, patients received 2 indacaterol 300 μg capsules. There was a washout period of 14-28 days between each treatment period. Patients received each treatment only once. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Indacaterol 300 μg; Drug: Placebo
- Indacaterol 150μg-indacaterol 600μg-placebo-indacaterol 300μg (Experimental): In treatment period 1, patients received 1 indacaterol 150 μg capsule + 1 placebo capsule; in treatment period 2, patients received 2 indacaterol 300 μg capsules; in treatment period 3, patients received 2 placebo capsules; and in treatment period 4, patients received 1 indacaterol 300 μg capsule + 1 placebo capsule. There was a washout period of 14-28 days between each treatment period. Patients received each treatment only once. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Indacaterol 300 μg; Drug: Placebo
- Indacaterol 300μg-placebo-indacaterol 600μg-indacaterol 150μg (Experimental): In treatment period 1, patients received 1 indacaterol 300 μg capsule + 1 placebo capsule; in treatment period 2, patients received 2 placebo capsules; in treatment period 3, patients received 2 indacaterol 300 μg capsules; and in treatment period 4, patients received 1 indacaterol 150 μg capsule + 1 placebo capsule. There was a washout period of 14-28 days between each treatment period. Patients received each treatment only once. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Indacaterol 300 μg; Drug: Placebo
- Indacaterol 600μg-indacaterol 300μg-indacaterol 150μg-placebo (Experimental): In treatment period 1, patients received 2 indacaterol 300 μg capsules; in treatment period 2, patients received 1 indacaterol 300 μg capsule + 1 placebo capsule; in treatment period 3, patients received 1 indacaterol 150 μg capsule + 1 placebo capsule; and in treatment period 4 patients received 2 placebo capsules. There was a washout period of 14-28 days between each treatment period. Patients received each treatment only once. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg; Drug: Indacaterol 300 μg; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol 150 μg was provided in powder filled capsules with a single dose dry powder inhaler (SDDPI).
Drug: Indacaterol 300 μg — Indacaterol 300 μg was provided in powder filled capsules with a single dose dry powder inhaler (SDDPI).
Drug: Placebo — Placebo to indacaterol was provided in powder filled capsules with a single dose dry powder inhaler (SDDPI).

SUMMARY:
The study was designed to obtain data about the efficacy and safety of 3 doses of indacaterol (150, 300, and 600 µg) in Japanese patients with chronic obstructive pulmonary disease (COPD) so that optimal dose(s) could be chosen for testing in later studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Japanese aged 40 to 75 years old
* Moderate to severe chronic obstructive pulmonary disease (COPD) with smoking history of at least 20 pack years

Exclusion Criteria:

* History of hospitalization for COPD exacerbation within past 6 months
* Use of long-term oxygen therapy
* History of asthma
* Respiratory tract infection within past 1 month
* Consistently very high or low blood sugar
* Clinically abnormal laboratory values or significant condition
* History of heart failure or heart attack within past 6 months
* History of long QT syndrome or long QT interval in electrocardiogram recorded at screening

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Principal Investigator — Novartis
Locations (8):
- Japan (8):
  - Novartis Investigative site, Kasukabe
  - Novartis Investigator Site, Kishiwada
  - Novartis Investigative Site, Kurume
  - Novartis Investigative Site, Obihiro
  - Novartis Investigative Site, Sagamihara
  - Novartis Investigative Site, Sapporo
  - Novartis Investigator Site, Tokyo
  - Novartis Investigative Site, Wakayama

REFERENCES:
- [Derived] Hosoe M, Woessner R, Matsushima S, Lawrence D, Kramer B. Efficacy, safety and pharmacokinetics of indacaterol in Caucasian and Japanese patients with chronic obstructive pulmonary disease: a comparison of data from two randomized, placebo-controlled studies. Clin Drug Investig. 2011;31(4):247-55. doi: 10.2165/11586520-000000000-00000. PMID 21184620

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Placebo-indacaterol 150μg-indacaterol 300μg-indacaterol 600μg | Indacaterol 150μg-indacaterol 600μg-placebo-indacaterol 300μg | Indacaterol 300μg-placebo-indacaterol 600μg-indacaterol 150μg | Indacaterol 600μg-indacaterol 300μg-indacaterol 150μg-placebo
Started | 12 | 13 | 11 | 14
Completed | 11 | 13 | 11 | 13
Not Completed | 1 | 0 | 0 | 1
Not completed — Subject withdrew consent | 1 | 0 | 0 | 0
Not completed — Subject no longer needs study drug | 0 | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Placebo-indacaterol 150μg-indacaterol 300μg-indacaterol 600μg | Indacaterol 150μg-indacaterol 600μg-placebo-indacaterol 300μg | Indacaterol 300μg-placebo-indacaterol 600μg-indacaterol 150μg | Indacaterol 600μg-indacaterol 300μg-indacaterol 150μg-placebo
Started | 11 | 13 | 11 | 13
Completed | 10 | 13 | 11 | 13
Not Completed | 1 | 0 | 0 | 0
Not completed — Subject withdrew consent | 1 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Placebo-indacaterol 150μg-indacaterol 300μg-indacaterol 600μg | Indacaterol 150μg-indacaterol 600μg-placebo-indacaterol 300μg | Indacaterol 300μg-placebo-indacaterol 600μg-indacaterol 150μg | Indacaterol 600μg-indacaterol 300μg-indacaterol 150μg-placebo
Started | 10 | 13 | 11 | 13
Completed | 10 | 13 | 11 | 11
Not Completed | 0 | 0 | 0 | 2
Not completed — Subject withdrew consent | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Treatment Period 4
Arm/Group | Placebo-indacaterol 150μg-indacaterol 300μg-indacaterol 600μg | Indacaterol 150μg-indacaterol 600μg-placebo-indacaterol 300μg | Indacaterol 300μg-placebo-indacaterol 600μg-indacaterol 150μg | Indacaterol 600μg-indacaterol 300μg-indacaterol 150μg-placebo
Started | 10 | 13 | 11 | 11
Completed | 10 | 13 | 11 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population included all 4 treatment groups who received indacaterol 150 µg, 300 µg, and 600 µg and placebo via a single dose dry powder inhaler (SDDPI) in 4 different sequences. Two capsules of study medication were inhaled in the morning between 8:00 and 10:00 am on Day 1 of each treatment period. Patients received each treatment only once. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 67.2 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 22 to 24 Hours Post-dose on Day 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made in each treatment period at 22, 23, and 24 hours post-dose on Day 2. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included patient, period, and treatment group as fixed effects and baseline FEV1 prior to drug administration in the treatment period as a covariate.
Time Frame: From 22 to 24 hours post-dose on Day 2
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug. Patients were included in the analysis if they had at least 1 FEV1 value at 22, 23, or 24 hours post-dose, and the data were not collected within 6 hours after the use of rescue medication.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol 600 μg: Two capsules of indacaterol 300 µg were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning between 8:00 and 10:00 am on Day 1 of the treatment period. Indacaterol 600 µg was administered only once to each patient. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Indacaterol 300 µg: One capsule of indacaterol 300 µg and 1 placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning between 8:00 and 10:00 am on Day 1 of the treatment period. Indacaterol 300 µg was administered only once to each patient. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Indacaterol 150 µg: One capsule of indacaterol 150 µg and 1 placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning between 8:00 and 10:00 am on Day 1 of the treatment period. Indacaterol 150 µg was administered only once to each patient. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Placebo: Two placebo capsules were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning between 8:00 and 10:00 am on Day 1 of the treatment period. Placebo was administered to each patient only once. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Indacaterol 600 μg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo
Number analyzed (Participants) | 47 | 47 | 47 | 46
Liters | 1.49 (0.010) | 1.48 (0.010) | 1.45 (0.010) | 1.33 (0.010)

2. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) From 5 Minutes to 4 Hours Post-dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made in each treatment period at 5, 15, and 30 minutes and 1, 2, and 4 hours post-dose on Day 1. The analysis included baseline FEV1 prior to drug administration in the treatment period as a covariate.
Time Frame: From 5 minutes to 4 hours post-dose on Day 1
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 600 μg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo
Number analyzed (Participants) | 48 | 47 | 48 | 47
Liters | 1.58 (0.009) | 1.57 (0.009) | 1.54 (0.009) | 1.42 (0.009)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) by Time Point From 5 Minutes to 12 Hours Post-dose on Day 1 and From 22 to 24 Hours Post-dose on Day 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made in each treatment period at 5, 15, and 30 minutes and 1, 2, 4, 8, and 12 hours on Day 1 and 22, 23, and 24 hours on Day 2. The analysis included baseline FEV1 prior to drug administration in the treatment period as a covariate.
Time Frame: From 5 minutes to 12 hours post-dose on Day 1 and from 22 to 24 hours post-dose on Day 2
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | Indacaterol 600 μg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo
Number analyzed (Participants) | 48 | 47 | 48 | 47
Liters
  5 minutes | 1.47 [1.45 to 1.48] | 1.48 [1.46 to 1.49] | 1.46 [1.45 to 1.48] | 1.36 [1.34 to 1.37]
  15 minutes | 1.50 [1.49 to 1.52] | 1.50 [1.48 to 1.51] | 1.49 [1.47 to 1.50] | 1.36 [1.34 to 1.37]
  30 minutes | 1.52 [1.50 to 1.54] | 1.52 [1.50 to 1.54] | 1.49 [1.47 to 1.51] | 1.35 [1.33 to 1.37]
  1 hour | 1.51 [1.49 to 1.53] | 1.51 [1.49 to 1.53] | 1.49 [1.47 to 1.51] | 1.36 [1.34 to 1.38]
  2 hours | 1.55 [1.53 to 1.57] | 1.54 [1.52 to 1.56] | 1.51 [1.49 to 1.53] | 1.36 [1.34 to 1.38]
  4 hours | 1.53 [1.50 to 1.55] | 1.53 [1.50 to 1.55] | 1.48 [1.46 to 1.50] | 1.35 [1.33 to 1.37]
  8 hour | 1.50 [1.48 to 1.52] | 1.51 [1.49 to 1.53] | 1.46 [1.44 to 1.48] | 1.30 [1.28 to 1.33]
  12 hours | 1.49 [1.47 to 1.51] | 1.47 [1.45 to 1.49] | 1.44 [1.42 to 1.46] | 1.30 [1.28 to 1.32]
  22 hours | 1.47 [1.45 to 1.49] | 1.46 [1.44 to 1.47] | 1.43 [1.41 to 1.45] | 1.29 [1.28 to 1.31]
  23 hours | 1.51 [1.49 to 1.53] | 1.49 [1.47 to 1.51] | 1.46 [1.44 to 1.48] | 1.33 [1.32 to 1.35]
  24 hours | 1.51 [1.49 to 1.52] | 1.50 [1.49 to 1.52] | 1.47 [1.45 to 1.49] | 1.35 [1.33 to 1.36]

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 5 Minutes to 12 Hours Post-dose on Day 1 and From 22 to 24 Hours Post-dose on Day 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made in each treatment period at 5, 15, and 30 minutes and 1, 2, 4, 8, and 12 hours on Day 1 and 22, 23, and 24 hours on Day 2. Standardized FEV1 AUC was calculated by the trapezoidal rule. The analysis included baseline FEV1 prior to drug administration in the treatment period as a covariate.
Time Frame: From 5 minutes to 12 hours post-dose on Day 1 and from 22 to 24 hours post-dose on Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 600 μg | Indacaterol 300 µg | Indacaterol 150 µg | Placebo
Number analyzed (Participants) | 47 | 46 | 47 | 45
Liters | 1.50 (0.009) | 1.49 (0.009) | 1.46 (0.009) | 1.32 (0.009)

ADVERSE EVENTS:
Groups:
- Indacaterol 150 μg: One capsule of indacaterol 150 µg and 1 placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning between 8:00 and 10:00 am on Day 1 of the treatment period. Indacaterol 150 µg was administered only once to each patient. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
- Indacaterol 300 μg: One capsule of indacaterol 300 µg and 1 placebo capsule were inhaled using a single dose dry powder inhaler (SDDPI) device in the morning between 8:00 and 10:00 am on Day 1 of the treatment period. Indacaterol 300 µg was administered only once to each patient. The short-acting β2-agonist salbutamol was available for rescue use throughout the study.
Arm/Group | Placebo | Indacaterol 150 μg | Indacaterol 300 μg | Indacaterol 600 μg
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/48 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 1/47 | 4/48 | 4/47 | 5/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | Indacaterol 150 μg (N=48) | Indacaterol 300 μg (N=47) | Indacaterol 600 μg (N=48)
SUBILEUS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | Indacaterol 150 μg (N=48) | Indacaterol 300 μg (N=47) | Indacaterol 600 μg (N=48)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.